CLINICAL TRIAL: NCT03238859
Title: 10 Days of Medial Prefrontal Cortex Theta Burst Stimulation (MPFC cTBS) as a Tool to Improve Clinical Outcomes and Decrease Frontal-striatal Reactivity to Cues Among Treatment-engaged Cocaine and Alcohol Users
Brief Title: 10 Days of Theta Burst Stimulation as a Tool to Treat Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Colleen A Hanlon, PhD, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00046438; R21DA041610 (NIH)
Record Dates: First submitted 2016-09-01; First posted 2017-08-03 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cocaine Dependence; Alcohol Dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real cTBS (Experimental): 10 days of real cTBS treatment will be given (3600 pulses to the left frontal pole as defined by EEG coordinate: FP1; 60 second pause after 1800 pulses; 110% RMT including a 30 second initial ramp period 80%-110% RMT; Magventure MagPro X100 Cool Coil).
  Interventions: Device: Real cTBS
- Sham cTBS (Sham Comparator): 10 days of sham cTBS treatment will be given (3600 pulses to the left frontal pole as defined by EEG coordinate: FP1; 60 second pause after 1800 pulses; 110% RMT including a 30 second initial ramp period 80%-110% RMT; Magventure MagPro X100 Cool Coil).
  Interventions: Device: Sham cTBS

INTERVENTIONS:
Device: Real cTBS — This will be delivered with the Magventure Magpro system; 3600 pulses with the active sham coil (double blinded using the USB key)
  Arms: Real cTBS
Device: Sham cTBS — This will be delivered with the sham Magventure Magpro system; 3600 pulses with the active sham coil (double blinded using the USB key)
  Arms: Sham cTBS

SUMMARY:
The goal of this double-blind sham controlled study is to evaluate the effeicacy of continuous theta burst stimulation to the frontal pole as a tool to decrease drug cue reactivity and improve treatment outcomes in treatment-engaged cocaine and alcohol users. All participants will be randomized to receive 10 days of real or sham rTMS to the frontal pole. Brain imaging data and behavioral assessments will be collected at 4 time points - before TMS, after 10 days of TMS, 1 month follow up and 2 month follow up.

DETAILED DESCRIPTION:
Cocaine dependence is a particularly difficult substance use disorder to treat. There is currently a lot of scientific inertia focused on the development of novel, neural circuit based strategies for intervention. A prior NARC funded pilot project in non-treatment seeking cocaine users demonstrated that a single session of medial prefrontal cortex theta burst stimulation (MPFC cTBS) decreases baseline frontal-striatal activity in limbic regions and decreases neural responses to cocaine uses. The effects of a single session however, erode over the first few hours after treatment. Sustainable effects require multiple days of treatment. GOAL: The next steps in pursuing this as a novel treatment are to 1) apply it to treatment-engaged patients and 2) determine whether several sessions of cTBS will produce sustainable and clinically-meaningful changes in cocaine use among these patients.

DESIGN: Treatment-engaged cocaine users and heavy alcohol users will be randomized to receive 10 sessions of real or sham LTD-like MPFC cTBS. This will be achieved by leveraging our existing partnership with the MUSC Center for Drug and Alcohol Programs (CDAP) and the Veterans Administration Substance Abuse Treatment Center Program (SATC) - which both provide a 4 week intensive outpatient treatment program. MPFC cTBS will be given during weeks 2 and 3 of the program. Functional MRI data and clinical assessments will be acquired during weeks 1, 4, and at participant's 1 month and 2 month Accountability/Continuity visits. Hypothesis: real cTBS treatment will enhance clinical outcomes (Aim 1 - including retention rates, number of clean urine drug screens during CDAP treatment, relapse rates at 1 and 2 months) and will produce a sustainable decrease in neural reactivity to cocaine cues (Aim 2 - week 1 versus week 4, 1 month & 2 month follow ups).

ELIGIBILITY:
Inclusion Criteria:

* Individuals from 21-65 years old currently enrolled in an intensive outpatient treatment program.

Exclusion Criteria:

* Participants will be excluded if they are not between 21-65 years old, have current or prior dependence (DSM-IV, because a DSM-V version of the SCID is not yet available) on prescription or psychoactive drugs other than cocaine, alcohol, or nicotine but including marijuana; past 6 month abuse of any prescription or psychoactive drugs excluding cocaine, marijuana, alcohol or nicotine, lifetime history of head injury with loss of consciousness, being pregnant or breast feeding, unstable medical illness (e.g., hypertension, diabetes, myocardial infarction), presence of ferromagnetic metal in their body, history of seizures. Additionally, to mitigate any potential risk of seizures. As mentioned above, all participants will receive the Clinical Institute Withdrawal Assessment of Alcohol (CIWAar) assessment before each TMS visit. Individuals with a CIWA score >5 will be excused from the study. All individuals with a history of medical detoxification or hospitalization for AUD (per the Assessments listed above), self-reported alcohol withdrawal seizures, or delirium tremens will be excluded from the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Drug cue reactivity | Baseline visit and 1 month follow up
  The effect of real versus sham cTBS on drug cue reactivity will be assessed by comparing the brain activity in the limbic system

SECONDARY OUTCOMES:
Number of Clean Urine Drug Screens | 1 month and 2 month follow up
  The effect of real versus sham cTBS on the number of clean urine drug screens will be assessed at the 1 and 2 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H Johnson Veterans Medical Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data is deidentified.